CLINICAL TRIAL: NCT01210339
Title: An Open-label, Randomized, Single-center, 2-way Cross-over Interaction Study, Evaluating the Effect of Esomeprazole 20 mg/Acetylsalicylic Acid 81 mg on the Pharmacodynamics and the Pharmacokinetics of Clopidogrel on Days 1 and 9 in Healthy Volunteers
Brief Title: An Interaction Study to Evaluate the Effect of Esomeprazole/Acetylsalicylic Acid on the Metabolism and Effect of Clopidogrel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D961FC00010
Record Dates: First submitted 2010-09-27; First posted 2010-09-28 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-10

CONDITIONS: Healthy Volunteers
Keywords: phase 1; cross-over; drug-drug Interaction; esomeprazole; acetylsalicylic acid; clopidogrel; healthy volunteers; cardiovascular disease; patients with acid associated gastrointestinal symptoms
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Treatment A (Clopidogrel 9 days), at least 14 days wash-out, Treatment B (Clopidogrel 4 days followed by Clopidogrel + Esomeprazole/ASA 5 days)
  Interventions: Drug: Clopidogrel; Drug: Esomeprazole/ASA
- 2 (Experimental): Treatment B (Clopidogrel 4 days followed by Clopidogrel + Esomeprazole/ASA 5 days), at least 14 days wash-out, Treatment A (Clopidogrel 9 days)
  Interventions: Drug: Clopidogrel; Drug: Esomeprazole/ASA

INTERVENTIONS:
Drug: Clopidogrel — Clopidogrel
Drug: Esomeprazole/ASA — 20 mg/81 mg once daily for five days (Day 5-9)
  Other Names: Axanum

SUMMARY:
The primary purpose of this study is to assess whether esomeprazole 20 mg/Acetyl Salicylic Acid (ASA) 81 mg affect the metabolism of clopidogrel.

ELIGIBILITY:
Inclusion Criteria:

* Male (aged between 18 and 45 years inclusive) or female (aged between 18 and 55 years inclusive) healthy volunteers
* Female healthy volunteers must be of non-childbearing potential or be of childbearing potential, be non-lactating and have a negative pregnancy test during the pre-entry visit and be using 1 clinically accepted method of contraception
* Have a body mass index between 19 and 30 kg/m2 inclusive
* No clinically significant abnormal findings at the physical examination as judged by the investigator

Exclusion Criteria:

* Any clinically significant abnormalities in laboratory screening results as judged by investigator
* Platelet count <150 x 10^9/L on Day -1 or any other conditions that would increase the risk of bleeding
* Previous bone marrow transplant
* Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2010-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
The effect of esomeprazole 20 mg/ acetylsalicylic acid 81 mg on the pharmacodynamics of clopidogrel by assessing maximal inhibition of platelet aggregation after 9 days of clopidogrel treatment relative to baseline | Pharmacodynamic sampling will be done before treatment period 1.
The effect of esomeprazole 20 mg/ acetylsalicylic acid 81 mg on the pharmacodynamics of clopidogrel by assessing maximal inhibition of platelet aggregation after 9 days of clopidogrel treatment relative to baseline | Pharmacodynamic sampling will be done after treatment period 1
The effect of esomeprazole 20 mg/ acetylsalicylic acid 81 mg on the pharmacodynamics of clopidogrel by assessing maximal inhibition of platelet aggregation after 9 days of clopidogrel treatment relative to baseline | Pharmacodynamic sampling will be done before treatment period 2.
The effect of esomeprazole 20 mg/ acetylsalicylic acid 81 mg on the pharmacodynamics of clopidogrel by assessing maximal inhibition of platelet aggregation after 9 days of clopidogrel treatment relative to baseline | Pharmacodynamic sampling will be done after treatment period 2.

SECONDARY OUTCOMES:
The effect of esomeprazole 20 mg/ acetylsalicylic acid 81 mg on the pharmacokinetics of the active metabolite of clopidogrel by assessing Area Under Curve (AUC) and Cmax.after 9 days of clopidogrel treatment | Pharmacokinetic sampling will be done at the end of treatment period 1 and 2 (Day 9).
The safety and tolerability of clopidogrel alone and in combination with esomeprazole/ acetylsalicylic acid | Safety will be monitored continuously. Adverse events will be collected from the first administration of Investigational Product (IP) throughout the study until the follow-up visit (on average) 7-10 days after last dose.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Nagy, MD, Study Director — AstraZeneca
Locations (1):
- Research Site, Uppsala, Sweden

REFERENCES:
- [Derived] Andersson T, Nagy P, Niazi M, Nylander S, Galbraith H, Ranjan S, Wallentin L. Effect of esomeprazole with/without acetylsalicylic acid, omeprazole and lansoprazole on pharmacokinetics and pharmacodynamics of clopidogrel in healthy volunteers. Am J Cardiovasc Drugs. 2014 Jun;14(3):217-27. doi: 10.1007/s40256-014-0073-4. PMID 24677117